CLINICAL TRIAL: NCT04291131
Title: Effects of Chronic Pain, Dyspnea, and Physical Activity Promotion on Functional Connectivity of the Brain in COPD
Brief Title: BRAIN, Symptoms, and Physical Activity in COPD
Acronym: BRAIN-SPA
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F3305-P
Record Dates: First submitted 2020-02-20; First posted 2020-03-02 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: COPD; Chronic Musculoskeletal Pain
Keywords: COPD; Pain; Dyspnea; Neuroimaging; Functional Connectivity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pain; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — None retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veterans with COPD: Veterans with COPD who will participate in a physical activity intervention or exercise program

SUMMARY:
Persons with COPD have both chronic musculoskeletal pain and dyspnea that require accurate diagnosis and treatment, ultimately to optimize functional status. The investigators propose to use advanced neuroimaging techniques to understand central mechanisms of chronic pain, dyspnea, and physical activity promotion in COPD. The investigators' novel proposal to correlate subjective symptoms (chronic pain and dyspnea) with an objective central biomarker (resting state functional connectivity) and examine their changes in response to a non-pharmacological, non-addictive physical activity intervention will personalize the care of Veterans with COPD.

DETAILED DESCRIPTION:
COPD is the nation's third leading cause of death and affects up to 11% of all VA healthcare patients. Patients with COPD experience significant dyspnea despite optimization of medical therapy. In addition, over half of patients with COPD experience chronic pain--largely musculoskeletal pain. Clinically, in patients who suffer from both chronic pain and dyspnea, it is difficult to distinguish a patient's perception of one symptom modulated by the other. Novel objective diagnostic tools are needed to complement patient self-report and accurately distinguish symptoms in patients who have both chronic pain and dyspnea to optimize clinical management. It is also important to study chronic pain and dyspnea in COPD because they are common barriers to engaging in physical activity (PA) and exercise. The clinical course of COPD is characterized by a downward spiral of dyspnea and chronic pain, physical inactivity, and significant functional limitation. Although chronic pain and dyspnea can be barriers, PA and exercise are powerful, but underused, non-addictive therapies for management of these symptoms in COPD. The investigators developed Every Step Counts (ESC), a technology-mediated intervention based on the Theory of Self-Regulation, to promote PA in COPD. The investigators have demonstrated ESC's safety, feasibility, and efficacy to increase PA and improve health-related quality of life in Veterans with COPD. In two separate studies using questionnaires, ESC has been shown to improve dyspnea in COPD and relieve chronic back pain in Veterans. An important next step is to understand the mechanisms of benefit of PA interventions, like ESC, in the many COPD patients with both chronic musculoskeletal pain and dyspnea to ultimately design better PA interventions and optimize treatment of these symptoms. Currently, the central mechanisms of chronic pain and dyspnea, and how they change in response to PA promotion in COPD are largely unknown. It has been shown that pre-stimulus resting state functional connectivity determines pain perception in healthy humans. Resting state fcMRI evaluates interactions between brain regions before a sensory event or when an explicit task is not being performed. These communications are altered in older adults with chronic musculoskeletal pain. Functional connectivity among regions specifically within the "default mode" network (DMN) (posterior cingulate, inferior parietal lobes, and medial frontal gyrus) have been examined in clinical disease states, as this network is reliably detected and well-characterized. Functional connectivity may be a novel biomarker of chronic pain and dyspnea.

Aim 1: Characterize and correlate the relationship between functional connectivity and chronic musculoskeletal pain and dyspnea in 30 persons with COPD (10 with both symptoms, 10 with chronic pain, and 10 with dyspnea).

Aim 2: Explore changes in functional connectivity and changes in symptoms in 30 persons with COPD after use of the ESC intervention to increase PA.

The investigators' proposed design will leverage enrollment of well-characterized participants with COPD already using the ESC PA intervention as part of a distinct and ongoing RR&D Merit Award. This proposal will provide insight into the biologically complex relationships between symptoms (chronic pain and dyspnea), behavior (PA), and biology at the central level (functional connectivity).

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 40 years of age
* Clinical diagnosis of COPD defined as either a ratio of FEV1 to forced vital capacity < 0.70 or chest CT evidence of emphysema or prior documentation of FEV1/FVC ratio of < 0.7 and clinical evidence of COPD (defined as 10 pack-year cigarette smoking history, dyspnea, or on bronchodilators)
* Will participate in a physical activity intervention or exercise program
* Competent to provide informed consent
* Willingness to make return visits and be available by telephone for duration of study

Exclusion Criteria:

* Female sex
* Claustrophobia
* History of seizures
* Known brain lesion
* Current diagnosis of bipolar disorder, schizophrenia, or psychotic disorder
* Cognitive disorder such as dementia
* Known metal in body including:

  * shrapnel
  * surgical medical clips
  * implants
  * pacemakers
  * metal-based tattoos

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with COPD
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn L. Moy, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Veterans With COPD
Started | 9
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Veterans With COPD
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Cortical thickness [Mean (Standard Deviation); unit: mm] | 2.24 (0.1)
Pain [Mean (Standard Deviation); unit: units on a scale] — Pain intensity will be measured with the Brief Pain Index. The Brief Pain Index rates pain intensity on a numbered scale of 0 - 10, with higher scores indicating more pain. Population: 6 participants did not complete questionnaire at baseline
  units on a scale
    number analyzed (Participants) | 3
    (all) | 4 (3)
Dyspnea [Mean (Standard Deviation); unit: units on a scale] — Dyspnea will be measured with the modified Medical Research Council scale from 0 to 4 where a higher score means greater dyspnea. Population: 1 missing value
  units on a scale
    number analyzed (Participants) | 8
    (all) | 2.38 (1.3)
Exercise capacity [Mean (Standard Deviation); unit: feet] — Population: Exercise capacity assessed by the 6-minute walk test where participant is asked to walk and cover as much ground as possible in 6 minutes. This is a validated test in patients with COPD.
  4 missing values
  feet
    number analyzed (Participants) | 5
    (all) | 1052 (263)
Physical Activity [Mean (Standard Deviation); unit: steps per day] — Population: 4 missing participants
  steps per day
    number analyzed (Participants) | 5
    (all) | 4519 (2497)

OUTCOME MEASURES:

1. Primary Outcome: Cortical Thickness
Description: Cortical thickness will be measured by brain MRIs that will assess functional connectivity and structural variables. Cortical thickness will be reported in millimeters.
Time Frame: 3 months
Population: Numbers do not match baseline numbers because of missing data. Participants may have completed only some assessments or did not have follow-up assessments.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Veterans With COPD
Number analyzed (Participants) | 6
mm | 2.2 (0.06)

2. Secondary Outcome: Exercise Capacity
Description: measured by the 6-minute walk test
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Veterans With COPD
Number analyzed (Participants) | 2
feet | 1410 (80)

3. Secondary Outcome: Physical Activity
Description: Measured by daily step counts
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Veterans With COPD
Number analyzed (Participants) | 5
steps per day | 4835 (3226)

4. Other Pre Specified Outcome: Pain Intensity
Description: Pain intensity will be measured with the Brief Pain Index. The Brief Pain Index rates pain intensity on a numbered scale of 0 - 10, with higher scores indicating more pain.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans With COPD
Number analyzed (Participants) | 2
units on a scale | 4 (1.41)

5. Other Pre Specified Outcome: Dyspnea
Description: Dyspnea will be measured with the modified Medical Research Council scale from 0 to 4 where a higher score means greater dyspnea.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans With COPD
Number analyzed (Participants) | 6
units on a scale | 1.83 (1.47)

ADVERSE EVENTS:
Time Frame: Duration of the study from enrollment to follow-up of approximately 3 months for each participant.
Arm/Group | Veterans With COPD
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Small sample size with missing data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT04291131/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT04291131/ICF_000.pdf